CLINICAL TRIAL: NCT05866614
Title: An Observational, Prospective Cohort Study to Evaluate Safety of Remsima® Subcutaneous in Patients With Rheumatoid Arthritis, Ankylosing Spondylitis, Psoriatic Arthritis and Psoriasis
Brief Title: A Study to Evaluate the Safety of Remsima® SC in the Treatment of RA, AS, PsA and Ps
Status: Recruiting | Type: Observational
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Other Study IDs: CT-P13 4.8
Record Dates: First submitted 2023-05-08; First posted 2023-05-19 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Rheumatoid Arthritis; Ankylosing Spondylitis; Psoriatic Arthritis; Psoriasis
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylitis, Ankylosing; Arthritis, Psoriatic; Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CT-P13 SC for RA patients: Patient will be treated as per the SmPC. The enrolled patient with RA will be administered Remsima® SC on the enrolment date and Remsima® SC injections will be continued according to the local standard of care. Study assessment will be done at least every 3 months through outpatient visit or telephone follow-up as part of routine care practice. Each outpatient visit is recommended to be done at least every 6 months and telephone follow-up will be done every 3 months after each outpatient visit to assess the patient.
  Interventions: Drug: Remsima SC
- CT-P13 SC for As, PsA and Ps patients: Patient will be treated as per the SmPC. The enrolled patient with AS, PsA, and Ps will be administered Remsima® SC on the enrolment date and Remsima® SC injections will be continued according to the local standard of care. Study assessment will be done at least every 3 months through outpatient visit or telephone follow-up as part of routine care practice. Each outpatient visit is recommended to be done at least every 6 months and telephone follow-up will be done every 3 months after each outpatient visit to assess the patient.
  Interventions: Drug: Remsima SC
- CT-P13 IV for As, PsA and Ps patients: Patient will be treated as per the SmPC. The enrolled patient with AS, PsA, and Ps will be administered Remsima® IV on the enrolment date and Remsima® IV infusions will be continued according to the local standard of care. Study assessment will be done at least every 3 months through outpatient visit or telephone follow-up as part of routine care practice. Each outpatient visit is recommended to be done at least every 6 months and telephone follow-up will be done every 3 months after each outpatient visit to assess the patient.
  Interventions: Drug: Remsima IV

INTERVENTIONS:
Drug: Remsima IV — Patient will be treated with Remsima IV as per the SmPC or
  Groups: CT-P13 IV for As, PsA and Ps patients
Drug: Remsima SC — Patient will be treated with Remsima SC as per the SmPC
  Groups: CT-P13 SC for As, PsA and Ps patients; CT-P13 SC for RA patients

SUMMARY:
This is an observational, prospective cohort study to evaluate the safety of Remsima® SC in the treatment of RA, AS, PsA and Ps.

DETAILED DESCRIPTION:
CT-P13(Remsima®) is an IgG1 chimeric human-murine mAb biosimilar to Remicade® (infliximab, Janssen Biologics B.V.) developed by CELLTRION, Inc.The purpose of this study is to assess the safety of Remsima® Subcutaneous (SC) in Rheumatoid Arthritis (RA), Ankylosing Spondylitis (AS), Psoriatic Arthritis (PsA) and Psoriasis (Ps) patients by evaluation of adverse events of special interest (AESI)

ELIGIBILITY:
Inclusion Criteria:

a.Patients with active RA having inadequate response to disease modifying antirheumatic drugs (DMARDs), including methotrexate (MTX) or b.Patients with severe, active and progressive RA not previously treated with MTX or other DMARDs c.Patients with severe, active AS who have responded inadequately to conventional therapy or d.Patients with active and progressive PsA when the response to previous DMARDs has been inadequate or e.Patients with moderate to severe plaque Ps who failed to respond to or who have a contraindication to, or are intolerant to other systemic therapy including cyclosporine, methotrexate or psoralen ultra-violet A.

* The Remsima® SC group will include all patients who meet one of the following classification at the time of enrolment:

  1. Biologic-naïve patients or
  2. Patients continuing on infliximab IV including Remsima® IV who will switch to Remsima® SC or
  3. Patients continuing on biologic treatments other than infliximab who will switch to Remsima® SC or
  4. Patients continuing on Remsima® SC (having commenced Remsima® SC treatment prior to enrolment)
* The Remsima® IV group will include all patients who meet one of the following classification at the time of enrolment:

  1. Biologic-naïve patients or
  2. Patients continuing on biologic treatments other than infliximab who will switch to Remsima® IV or
  3. Patients continuing on infliximab IV including Remsima® IV who will switch to or maintain Remsima® IV * Note: Switching from Remsima® SC to Remsima® IV is not allowed.

Exclusion Criteria:

1. Patients with a history of hypersensitivity to murine, chimeric, human, or humanized proteins or any of the excipients of Remsima® SC or Remsima® IV, whichever the patients are going to be treated in each treatment group, listed in the Summary of Product Characteristics (SmPC) of each product.
2. Patients with any reported contraindications for Remsima® SC or Remsima® IV according to the SmPC of each product.

   1. Patients with active tuberculosis (TB)
   2. Patients with inactive (latent) TB who are not willing or not compliant with TB prophylaxis or a past diagnosis of TB without sufficient documentation of complete resolution following treatment.
   3. Patients with severe infection such as sepsis, abscesses and opportunistic infections (including, disseminated herpes simplex virus, candidiasis but not limited to)
   4. Patients with a current or past history of chronic infection with human immunodeficiency virus (HIV), hepatitis B and hepatitis C
   5. Patients with moderate or severe heart failure (New York Heart Association [NYHA] class III/IV)
   6. Patients for whom there are investigator concerns about treatment with tumour necrosis factor alpha (TNF-α) inhibitor, such as a history of any malignancy within the previous five years prior to enrolment, may be excluded at the investigator's discretion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female patients with RA will be enrolled and treated with Remsima® SC. Male or female patients with AS, PsA, and Ps will be enrolled and treated with either Remsima® SC or Remsima® IV. Patients will be considered for enrolment in the study if they meet all of the inclusion criteria and none of the exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 864 (Estimated)
Dates: Start 2023-01-13 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
evaluation of adverse events of special interest (AESI) | through study completion, an average of 2 years
  The safety population will consist of all patients who receive at least 1 (full or partial) dose of either Remsima® SC or Remsima® IV during study period. Analyses will be performed on the observed cases. All safety data will be summarized by treatment groups as appropriate in the Safety population.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Purpan Hôpital Pierre Paul Riquet, Toulouse, France